CLINICAL TRIAL: NCT05524194
Title: A Phase I/II, Multicenter, Open-Label, Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Pharmacodynamics of 6MW3511 in Patients With Advanced Solid Tumor
Brief Title: 6MW3511 in Patients With Advanced Solid Tumor
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6MW3511-2022-CP101
Record Dates: First submitted 2022-08-28; First posted 2022-09-01 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Solid Tumors
MeSH Terms: interventions — Infusions, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: 6MW3511 (Experimental): Subjects will receive 6MW3511 by intravenous administration.
  Interventions: Drug: Intravenous Infusion

INTERVENTIONS:
Drug: Intravenous Infusion — Dose-limiting toxicity (DLT) are assessed during the first 3 weeks (21 days) after initial administration. Then, the intended dosing frequency is every 2 weeks (Q2W).

SUMMARY:
This is a phase I/II , open-label, multicenter single arm study designed to evaluate the safety, tolerability, pharmacokinetic (PK), and immunogenicity of 6MW3511.

DETAILED DESCRIPTION:
This is a Phase I/II, open-label, dose-escalation trial with consecutive parallel-group expansion in selected solid tumor indications. The study consists of a dose escalation phase to determine the maximum tolerated dose (MTD), or recommended Phase 2 dose (RP2D) for 6MW3511, and a dose expansion phase which will characterize treatment of 6MW3511 at the RP2D.

ELIGIBILITY:
Inclusion Criteria:

1. In dose-escalation cohorts, histologically or cytologically documented advanced or metastatic solid tumor that is refractory/relapsed to standard therapies, or for which no effective standard therapy is available, or the subject refuses standard therapy.In the dose-expansion cohorts , histologically or cytologically confirmed selected advanced solid tumors (to be determined).
2. Male or female subjects aged over 18 years old (inclusive) and not more than 80 years old (inclusive).
3. Eastern Cooperative Oncology Group (ECOG) Performance Score of 0 or 1.

Exclusion Criteria:

1. History of other malignant tumors within 3 years, except for the tumors that had been cured.
2. Symptomatic or active central nervous system metastasis.
3. Patients with active autoimmune disease.
4. History of allogeneic hematopoietic stem cell transplantation or organ transplantation.
5. Patients previously treated with PD-（L）1/ TGF-β antibody or combined PD-（L）1 with TGF-β antibody.
6. Pregnant or breast feeding.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a Dose Limiting Toxicity (DLT) | Up to Week 3
  DLTs will be assessed during the first 3 weeks of treatment for dose-escalation phase.
Number of participants with adverse events (AEs) | Up to 4 weeks after last treatment
  Characterization of incidence, severity and abnormal clinically significant laboratory findings of AEs.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1.
Disease control rate (DCR) | Up to 2 years
  The DCR is defined as the proportion of subjects with CR, PR, or SD (subjects achieving SD will be included in the DCR if they maintain SD for ≥8 weeks) based on RECIST Version 1.1.
Maximum observed concentration (Cmax) of 6MW3511 | Up to 4 weeks after last treatment
  The endpoints for assessment of PK of 6MW3511 include serum concentrations of 6MW3511 at different timepoints after administration.
Number of subjects who develop detectable anti-drug antibodies (ADAs) | Up to 4 weeks after last treatment
  The immunogenicity of 6MW3511 will be assessed by summarizing the number of subjects who develop detectable anti-drug antibodies (ADAs).